CLINICAL TRIAL: NCT06528392
Title: Efgartigimod for Stiff Person Syndrome (ESPS)
Acronym: ESPS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY006922
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stiff-Person Syndrome
Keywords: Stiff-Person Syndrome; Efgartigimod
MeSH Terms: conditions — Stiff-Person Syndrome | interventions — efgartigimod alfa

STUDY DESIGN:
Intervention Model Description: This is an exploratory, single arm treatment, non-inferiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- subcutaneous Efgartigimod-hyaluronidase (EFG) (Experimental): Participants with GAD65-antibody positive SPS will be given subcutaneous Efgartigimod-hyaluronidase (EFG).
  Interventions: Biological: Efgartigimod

INTERVENTIONS:
Biological: Efgartigimod — Efgartigiomd-hyaluroidase (EFG) is a neonatal Fc receptor (FcRn) inhibitor, which blocks the recycling of Immunoglobulin G (IgG), including pathogenic IgG

SUMMARY:
The goal of this clinical trial is to examine the proportion of patients with stiff person syndrome with no worsening in stiffness and/or spasms while on efgartigimod-hyaluronidase (EFD) when compared to their current treatment. The main questions it aims to answer are:

* proportion of patients with stiff person syndrome with no worsening in DSI and HSS scores
* whether there are changes in laboratory values, vital signs, electrocardiogram, or depression, and suicide risk during the trial, as well as the incidence of any adverse events.

Participants will come to the clinic up to 18 times and have up to 5 phone call visits during the course of the trial. During these visits a variety of measures will be collected, including blood samples, neurological and physical exams, patient reported outcomes on stiffness, spasms, depression, and suicide risk.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80, men and women, capable of giving informed consent.
2. Must have unexplained stiffness of limb and axial (trunk) muscles and involuntary striated muscle spasms.
3. DSI and HHS must be >=2 (to allow for detection of improvement).
4. Presence of serum (or CSF) anti-GAD antibodies regardless of titers.
5. Stable dosage for at least two months before screening visit with antispasmodics (muscle relaxants, benzodiazepines, baclofen).
6. Women with children bearing potential must be willing to use highly effective contraception method during and for a minimum of 90 days after the last dose of IP.

Exclusion Criteria:

1. Exclusionary conditions:

1a. type 1 DM

1b. Cancer, except basal cell skin cancer

1c. Infections: HIV, Hepatitis B or C, clinically significant active infection not sufficiently resolved in the investigator's opinion

1d. Serum IgG (<6 g/L) at screening

1e. pregnancy/breast feeding. 2. Exclusionary medications: rituximab within 6 months of screening. 3. IVIG or PLEX treatment 4 weeks prior to screening. 4. History of any type of solid organ or bone marrow transplant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of Stiffness Index (DSI) | From enrollment to the end of treatment at week 13
  DSI is a validated indicator or stiffness. Scores range from 0 to 6 and reflect the extent of stiffness. One point is given for stiffness in each of the following areas: lower trunk, upper trunk, legs, arms, face and abdomen.
heightened sensitivity score (HSS) | From enrollment to end of treatment at week 13
  HSS measures changes in the frequency of spasms. Scores range from 1 to 7; one point given for each source or type of spasm: unexpected noises, visual stimuli, somatosensory stimuli, voluntary activities, emotional upset or stress, no specific stimuli, or nocturnal spasms.

SECONDARY OUTCOMES:
Proportion of patients with SPS who are treatment responders | enrollment to end of 13 weeks
  Proportion of patients with SPS who are treatment responders, defined as: >= 2 points reduction in the distribution of stiffness index (DSI) AND >= 1 point reduction in heightened sensitivity score (HSS)
The duration of time patients maintain responder status | from enrollment to end of treatment at week 13
  A responder is defined as one having >= 2 points reduction in the distribution of stiffness index (DSI) AND >= 1 point reduction in heightened sensitivity score (HSS)
Modified Rankin Scale | From enrollment to end of treatment at week 13

CONTACTS AND LOCATIONS:
Overall Officials: Tuan H Vu, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared between designated study sites during the trial. After the end of the trial data may be shared but this has yet to be determined.